CLINICAL TRIAL: NCT01497158
Title: Promoting Home Smoking Restrictions: Biomarker Feedback to Cohabitating Smoking and Non-Smoking Adults
Brief Title: Promoting Home Smoking Restrictions: Biomarker Feedback to Smoking and Non-Smoking Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007NT053
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Smoking Cessation; Tobacco Use Disorder
Keywords: tobacco cessation
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Participants who received only self-help brochure regarding environmental tobacco smoking (ETS) exposure in the home.
  Interventions: Other: Self-help brochure
- Active Group (Active Comparator): Participants who received self-help brochure regarding environmental tobacco smoking (ETS) exposure in the home and biomarker feedback from the urine of cohabitating adult non-smoker in the home.
  Interventions: Other: Self-help brochure; Other: Biomarker feedback

INTERVENTIONS:
Other: Self-help brochure — Self help brochure given at baseline visit.
Other: Biomarker feedback — Biomarker feedback from urine of adult non-smoker in the home.
  Arms: Active Group

SUMMARY:
This study is directed at decreasing home environmental tobacco smoking (ETS) exposure with a novel approach of adoption of home smoking restrictions. This will be done by providing the cohabitating smoker and non-smoker with biomarker feedback documenting exposure to ETS. The intent is to identify an intervention strategy(ies) to reduce ETS exposure.

DETAILED DESCRIPTION:
This is a two-group interventional trial targeting cohabitating smokers and non-smokers. Participants will be randomized to the control condition or biomarker feedback group.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Cohabitating Non-Smoker (control) and smoker (active)
* Smoker must test > 6ppm on carbon dioxide (CO) test and non-smoker < 6ppm
* General good health
* Written informed consent
* Live within Twin Cities 7 county metropolitan area (Minnesota)
* Plan to live in same home for 6 months and be willing for researchers to come to their home

Exclusion Criteria:

* Individuals that live in a treatment facility or shelter
* Individuals endorsing current domestic violence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Comparison of Self-Reported Home Smoking Restrictions - Active Counseling | From baseline to week 12
  Received self-help brochure and biomarker feedback from urine collected from non-smoking adult in home. Outcome criteria categorized into 3 areas: establishment of a complete ban (defined as no one allowed to smoke anywhere, ever), some restrictions (smoking allowed in some places or some time), and no restrictions (smoking permitted anywhere, no rules).
Comparison of Self-Reported Home Smoking Restrictions - Control Group | From baseline to week 12
  Received only self-help brochure on home ETS exposure. Outcome criteria categorized into 3 areas: establishment of a complete ban (defined as no one allowed to smoke anywhere, ever), some restrictions (smoking allowed in some places or some time), and no restrictions (smoking permitted anywhere, no rules).

CONTACTS AND LOCATIONS:
Overall Officials: Janet Thomas, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States